CLINICAL TRIAL: NCT04640571
Title: Impact of Metformin and Polysorbate 80 on Drug Absorption and Disposition
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Responsible Party: Principal Investigator, James E Polli, Professor, University of Maryland, Baltimore
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: HP-00090086
Record Dates: First submitted 2020-11-09; First posted 2020-11-23 (Actual); Results first posted 2024-07-16 (Actual); Last update posted 2024-07-16 (Actual); Status verified 2024-07

CONDITIONS: Bile Salt Export Pump (BSEP) Transporter; Polysorbate 80
Keywords: healthy volunteer; pharmacokinetics; excipient; transporter
MeSH Terms: conditions — Cholestasis, progressive familial intrahepatic 2 | interventions — Pravastatin; Chenodeoxycholic Acid; Valacyclovir; Enalaprilat

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (6):
- placebo, then metformin, then polysorbate 80 (Experimental): Placebo is one twice a day, metformin is 500mg twice a day, and polysorbate 80 is 400mg twice a day
  Interventions: Drug: pravastatin and chenodeoxycholic acid, after metformin and placebo; Drug: valacyclovir, chenodeoxycholic acid, and enalaprilat, after polysorbate 80 and placebo
- metformin, then polysorbate 80, then placebo (Experimental): Placebo is one twice a day, metformin is 500mg twice a day, and polysorbate 80 is 400mg twice a day
  Interventions: Drug: pravastatin and chenodeoxycholic acid, after metformin and placebo; Drug: valacyclovir, chenodeoxycholic acid, and enalaprilat, after polysorbate 80 and placebo
- polysorbate 80, then placebo, then metformin (Experimental): Placebo is one twice a day, metformin is 500mg twice a day, and polysorbate 80 is 400mg twice a day
  Interventions: Drug: pravastatin and chenodeoxycholic acid, after metformin and placebo; Drug: valacyclovir, chenodeoxycholic acid, and enalaprilat, after polysorbate 80 and placebo
- polysorbate 80, then metformin, then placebo (Experimental): Placebo is one twice a day, metformin is 500mg twice a day, and polysorbate 80 is 400mg twice a day
  Interventions: Drug: pravastatin and chenodeoxycholic acid, after metformin and placebo; Drug: valacyclovir, chenodeoxycholic acid, and enalaprilat, after polysorbate 80 and placebo
- placebo, then polysorbate 80, then metformin (Experimental): Placebo is one twice a day, metformin is 500mg twice a day, and polysorbate 80 is 400mg twice a day
  Interventions: Drug: pravastatin and chenodeoxycholic acid, after metformin and placebo; Drug: valacyclovir, chenodeoxycholic acid, and enalaprilat, after polysorbate 80 and placebo
- metformin, then placebo, then polysorbate 80 (Experimental): Placebo is one twice a day, metformin is 500mg twice a day, and polysorbate 80 is 400mg twice a day
  Interventions: Drug: pravastatin and chenodeoxycholic acid, after metformin and placebo; Drug: valacyclovir, chenodeoxycholic acid, and enalaprilat, after polysorbate 80 and placebo

INTERVENTIONS:
Drug: pravastatin and chenodeoxycholic acid, after metformin and placebo — single oral dose of pravastatin 80 mg and chenodeoxycholic acid 250 mg
Drug: valacyclovir, chenodeoxycholic acid, and enalaprilat, after polysorbate 80 and placebo — single oral dose of valacyclovir 500 mg, chenodeoxycholic acid 250 mg, and enalaprilat 20 mg

SUMMARY:
The study employs two-sub-studies that share a common placebo arm.

The objective of one sub-study is to assess the impact of metformin on pravastatin and chenodeoxycholic acid pharmacokinetics. We hypothesize that metformin represses the bile salt export pump (BSEP) in the liver, which excretes pravastatin and chenodeoxycholic acid from the liver into the bile.

The objective of the other sub-study is to assess the impact of polysorbate 80 on valacyclovir, chenodeoxycholic acid, and enalaprilat pharmacokinetics. We hypothesize that polysorbate 80 inhibits uptake transporters in the intestine, which absorb valacyclovir and chenodeoxycholic acid in the gut via the peptide transporter 1 (PepT1) and apical sodium-bile acid transporter (ASBT), respectively. Enalaprilat is passively absorbed but with low permeability, and thus serves as a passive absorption reference.

ELIGIBILITY:
Inclusion Criteria:

* Subject is healthy, as determined by screening evaluation that is not greater than 60 days before the first study visit.
* Subject is male or female between 18 and 65 years of age, inclusive.
* Subject is an acceptable candidate for venipuncture.
* Subject is willing to stop all non-routine OTC medications, as well as vitamins, dietary supplements, and herbals, for 24 hours prior to study drug administration and during pharmacokinetic study visits.

Exclusion Criteria:

* Subject has a significant medical disease (including cardiovascular, pulmonary, hematologic, endocrine, immunologic, neurologic, renal, gastrointestinal, metabolic, or psychiatric).
* Subject has a clinically significant history or presence of any clinically significant gastrointestinal pathology (e.g. chronic diarrhea, inflammatory bowel diseases), unresolved gastrointestinal symptoms (e.g. diarrhea, vomiting), liver or kidney disease, or other conditions known to interfere with the absorption, distribution, metabolism or excretion of study drugs.
* Subject has a history of liver or gallbladder disease, or history of myopathy
* Subject has a history of angioedema either with or without previous treatment with an angiotensin converting enzyme inhibitor.
* Subject was previously diagnosed with diabetes, or treated with antidiabetic agents
* Subject has a history of alcohol or drug abuse, which in the opinion of the PI or medical physician, could jeopardize the subject's health or would compromise the subject's ability to participate in this trial.
* Subject is pregnant, breast feeding, or trying to become pregnant.
* Female subject of childbearing potential is unwilling or unable to use a medically acceptable method of contraception throughout the entire study period and for one week after the study is completed. Medically acceptable methods of contraception that may be used by the subject and/or her partner are: oral birth control pill, condom with spermicide, diaphragm with spermicide, IUD, vaginal spermicidal suppository, surgical sterilization of patient or their partner(s), abstinence, or hormonal-based patches, ring, injections, and implants.
* Subject routinely uses (i.e. daily or weekly) prescription medication except hormonal birth control medication, routinely uses (i.e. daily or weekly) OTC medication, or routinely uses niacin to treat hypercholesterolemia. OTC medications do not include vitamins, dietary supplements, or herbals.
* Subject routinely uses (i.e. daily or weekly) acid blockers, antacids, anti-diarrhea, stimulants, appetite suppressants, or anti-nausea medication or other drugs that modulate GI function.
* Subject is currently taking metformin, valacyclovir, acyclovir, chenodiol, pravastatin, enalapril, enalaprilat, or medications known to interact with any of these medications.
* Subject has a history or allergy or sensitivity to metformin, valacyclovir, acyclovir, chenodiol, pravastatin, polysorbate 80, enalapril, enalaprilat, or history of any drug hypersensitivity or intolerance which, in the opinion of the PI or medical physician, would compromise the safety of the subject or the study.
* Subject has liver impairment as assessed by alanine aminotransferase (ALT), aspartate aminotransferase (AST), or total bilirubin levels greater than the upper limit of normal (ULN).
* Subject has renal impairment as assessed by creatinine clearance lower than 60mL/min/1.73m2, using the CKDEPI formula.
* Subject is not willing or able to be adherent to study protocol (e.g., study visits).
* Subject has a condition in which in the opinion of the PI or medical physician would increase risk to the subject or interfere with the integrity of the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2021-11-01 (Actual); Study Completion 2021-11-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Maryland, Baltimore, Maryland, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: UMB IRB, a subject is enrolled if they signed a consent form, regardless if they passed screening.
Period: Overall Study
Arm/Group | Placebo, Then Metformin, Then Polysorbate 80 | Metformin, Then Polysorbate 80, Then Placebo | Polysorbate 80, Then Placebo, Then Metformin | Polysorbate 80, Then Metformin, Then Placebo | Placebo, Then Polysorbate 80, Then Metformin | Metformin, Then Placebo, Then Polysorbate 80
Started | 2 | 2 | 2 | 2 | 2 | 4
Completed | 2 | 2 | 2 | 2 | 2 | 2
Not Completed | 0 | 0 | 0 | 0 | 0 | 2
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Population: Dropped participants did not contribute to the analysis.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo, Then Metformin, Then Polysorbate 80 | Metformin, Then Polysorbate 80, Then Placebo | Polysorbate 80, Then Placebo, Then Metformin | Polysorbate 80, Then Metformin, Then Placebo | Placebo, Then Polysorbate 80, Then Metformin | Metformin, Then Placebo, Then Polysorbate 80 | Total
Number analyzed (Participants) | 2 | 2 | 2 | 2 | 2 | 2 | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 2 | 2 | 2 | 2 | 2 | 2 | 12
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Full Range); unit: years] | 28.5 [26 to 31] | 26.5 [23 to 30] | 28.5 [28 to 29] | 26.5 [24 to 29] | 40 [28 to 52] | 28 [24 to 32] | 29.7 [23 to 52]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 0 | 1 | 1 | 1 | 7
  Male | 0 | 0 | 2 | 1 | 1 | 1 | 5
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White/Caucasian | 2 | 1 | 0 | 0 | 1 | 0 | 4
  Black/African American | 0 | 0 | 1 | 2 | 1 | 2 | 6
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 1 | 0 | 0 | 0 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 2 | 2 | 2 | 2 | 2 | 2 | 12

OUTCOME MEASURES:

1. Primary Outcome: Area-Under-the-Curve (AUC) of Pravastatin After Metformin
Description: Pravastatin AUC after metformin, compared to pravastatin AUC after placebo. AUC units are concentration x time (i.e. ng/ml x h).
Time Frame: 0-10 hours
Measure: Mean (Standard Error); unit: ng/ml × h
Groups:
- Metformin: Participants took 500 mg metformin b.i.d. for 6 days. On day 7, participants were administered 80 mg pravastatin and 250 mg chenodeoxycholic acid.
- Placebo: Participants took one placebo b.i.d. for 6 days. On day 7, participants were administered 500 mg valacyclovir, 250 mg CDCA, 20 mg enalaprilat, and 80 mg pravastatin.
Arm/Group | Metformin | Placebo
Number analyzed (Participants) | 12 | 12
ng/ml × h | 264.2 (34.1) | 170.5 (24.7)
Statistical Analysis 1: Comparison: Metformin vs Placebo; Test type: Equivalence — Simple one-way t-test to assess if pravastatin AUC value is larger after metformin than after placebo; p = 0.02, t-test, 1 sided

2. Primary Outcome: Peak Plasma Concentration (Cmax) of Pravastatin After Metformin
Description: Pravastatin Cmax after metformin, compared to pravastatin Cmax after placebo. Cmax units are concentration (i.e. ng/ml).
Time Frame: 0-10 hours
Measure: Mean (Standard Error); unit: ng/ml
Groups:
- Placebo: Participants took one placebo b.i.d. for 6 days. On day 7, participants were administered 500 mg valacyclovir, 250 mg chenodeoxycholic acid, 20 mg enalaprilat, and 80 mg pravastatin.
Arm/Group | Metformin | Placebo
Number analyzed (Participants) | 12 | 12
ng/ml | 119.3 (17.7) | 86.43 (15.86)
Statistical Analysis 1: Comparison: Metformin vs Placebo; Test type: Equivalence — Simple one-way t-test to assess if pravastatin Cmax value is larger after metformin than after placebo; p < 0.05, t-test, 1 sided

3. Primary Outcome: Area-Under-the-Curve (AUC) of Chenodeoxycholic Acid After Metformin
Description: Baseline-corrected chenodeoxycholic acid AUC after metformin. AUC Units are concentration x time (i.e. ng/ml x h). Baseline-corrected chenodeoxycholic acid is chenodeoxycholic acid concentration minus chenodeoxycholic acid concentration value at time zero (i.e. t=0).
Time Frame: 0-10 hours
Measure: Mean (Standard Error); unit: ng/ml x h
Arm/Group | Metformin | Placebo
Number analyzed (Participants) | 12 | 12
ng/ml x h | 4646 (352) | 4665 (370)
Statistical Analysis 1: Comparison: Metformin vs Placebo; Test type: Equivalence — Simple one-way t-test to assess if CDCA AUC value is reduced after metformin than after placebo; p < 0.05, t-test, 1 sided

4. Primary Outcome: Peak Plasma Concentration (Cmax) of Chenodeoxycholic Acid After Metformin
Description: Baseline-corrected chenodeoxycholic acid Cmax after metformin. Cmax units are concentration (i.e. ng/ml). Baseline-corrected chenodeoxycholic acid is chenodeoxycholic acid concentration minus chenodeoxycholic acid concentration value at time zero (i.e. t=0).
Time Frame: 0-10 hours
Measure: Mean (Standard Error); unit: ng/ml
Arm/Group | Metformin | Placebo
Number analyzed (Participants) | 12 | 12
ng/ml | 2695 (453) | 2881 (351)
Statistical Analysis 1: Comparison: Metformin vs Placebo; Test type: Equivalence — Simple one-way t-test to assess if CDCA Cmax value is reduced after metformin than after placebo; p < 0.05, t-test, 1 sided

5. Primary Outcome: Area-Under-the-Curve (AUC) of Acyclovir After Polysorbate 80
Description: Acyclovir AUC after polysorbate 80. AUC units are concentration x time (i.e. ng/ml x h).
Time Frame: 0-10 hours
Measure: Mean (Standard Error); unit: ng/ml x h
Groups:
- Polysorbate 80: Participants took 400 mg polysorbate 80 b.i.d. for 6 days. On day 7, participants were administered 500 mg valacyclovir, 250 mg chenodeoxycholic acid, 20 mg enalaprilat, and 400 mg polysorbate 80.
Arm/Group | Polysorbate 80 | Placebo
Number analyzed (Participants) | 12 | 12
ng/ml x h | 10039 (903) | 9839 (782)
Statistical Analysis 1: Comparison: Polysorbate 80 vs Placebo; Test type: Equivalence — Simple one-way t-test to assess if acyclovir AUC value is reduced after polysorbate 80 than after placebo; p < 0.05, t-test, 1 sided

6. Primary Outcome: Peak Plasma Concentration (Cmax) of Acyclovir After Polysorbate 80
Description: Acyclovir Cmax after polysorbate 80. Cmax units are concentration (i.e. ng/ml).
Time Frame: 0-10 hours
Measure: Mean (Standard Error); unit: ng/ml
Arm/Group | Polysorbate 80 | Placebo
Number analyzed (Participants) | 12 | 12
ng/ml | 3363 (348) | 3230 (367)
Statistical Analysis 1: Comparison: Polysorbate 80 vs Placebo; Test type: Equivalence — Simple one-way t-test to assess if acyclovir Cmax value is reduced after polysorbate 80 than after placebo; p < 0.05, t-test, 1 sided

7. Primary Outcome: Area-Under-the-Curve (AUC) of Chenodeoxycholic Acid (CDCA) After Polysorbate 80
Description: Baseline-corrected Chenodeoxycholic acid AUC after polysorbate 80. AUC units are concentration x time (i.e. ng/ml x h). Baseline-corrected chenodeoxycholic acid is chenodeoxycholic acid concentration minus chenodeoxycholic acid concentration value at time zero (i.e. t=0).
Time Frame: 0-10 hours
Measure: Mean (Standard Error); unit: ng/ml x h
Arm/Group | Polysorbate 80 | Placebo
Number analyzed (Participants) | 12 | 12
ng/ml x h | 4964 (300) | 4665 (370)
Statistical Analysis 1: Comparison: Polysorbate 80 vs Placebo; Test type: Equivalence — Simple one-way t-test to assess if CDCA AUC value is reduced after polysorbate 80 than after placebo; p < 0.05, t-test, 1 sided

8. Primary Outcome: Peak Plasma Concentration (Cmax) of Chenodeoxycholic Acid (CDCA) After Polysorbate 80
Description: Baseline-corrected Chenodeoxycholic acid Cmax after polysorbate 80. Cmax units are concentration (i.e. ng/ml). Baseline-corrected chenodeoxycholic acid is chenodeoxycholic acid concentration minus chenodeoxycholic acid concentration value at time zero (i.e. t=0).
Time Frame: 0-10 hours
Measure: Mean (Standard Error); unit: ng/ml
Arm/Group | Polysorbate 80 | Placebo
Number analyzed (Participants) | 12 | 12
ng/ml | 2960 (276) | 2881 (351)
Statistical Analysis 1: Comparison: Polysorbate 80 vs Placebo; Test type: Equivalence — Simple one-way t-test to assess if CDCA Cmax value is reduced after polysorbate 80 than after placebo; p < 0.05, t-test, 1 sided

9. Primary Outcome: Area-Under-the-Curve (AUC) of Enalaprilat After Polysorbate 80
Description: Enalaprilat AUC after polysorbate 80. AUC units are concentration x time (i.e. ng/ml x h).
Time Frame: 0-10 hours
Measure: Mean (Standard Error); unit: ng/ml x h
Arm/Group | Polysorbate 80 | Placebo
Number analyzed (Participants) | 12 | 12
ng/ml x h | 10.98 (3.05) | 12.10 (2.71)
Statistical Analysis 1: Comparison: Polysorbate 80 vs Placebo; Test type: Equivalence — Simple one-way t-test to assess if enalaprilat AUC value is increased after polysorbate 80 than after placebo; p < 0.05, t-test, 1 sided

10. Primary Outcome: Peak Plasma Concentration (Cmax) of Enalaprilat After Polysorbate 80
Description: Enalaprilat Cmax after polysorbate 80. Cmax units are concentration (i.e. ng/ml).
Time Frame: 0-10 hours
Measure: Mean (Standard Error); unit: ng/ml
Arm/Group | Polysorbate 80 | Placebo
Number analyzed (Participants) | 12 | 12
ng/ml | 1.720 (0.480) | 2.080 (0.540)
Statistical Analysis 1: Comparison: Polysorbate 80 vs Placebo; Test type: Equivalence — Simple one-way t-test to assess if enalaprilat Cmax value is increased after polysorbate 80 than after placebo; p < 0.05, t-test, 1 sided

11. Secondary Outcome: Area-Under-the-Curve (AUC) of Endogenous Bile Acids After Polysorbate 80
Description: For each of 15 endogenous bile acid, endogenous bile acid AUC after polysorbate 80, compared to endogenous bile acid AUC after placebo. AUC units are concentration x time (i.e. ng/ml x h).
Time Frame: 0-10 hours
Measure: Mean (Standard Error); unit: ng/ml x h
Arm/Group | Polysorbate 80 | Placebo
Number analyzed (Participants) | 12 | 12
ng/ml x h
  Cholic acid | 264.3 (50.6) | 259.7 (64.6)
  Glycocholic acid | 1171 (185) | 1053 (187)
  Taurocholic acid | 280.8 (40.9) | 248.1 (39.5)
  Deoxycholic acid | 1451 (242) | 1222 (158)
  Glycodeoxycholic acid | 1655 (183) | 1507 (200)
  Taurodeoxycholic acid | 346.7 (38.6) | 329.3 (53.1)
  Chenodeoxycholic acid | 5718 (409) | 5552 (471)
  Glycochenodeoxycholic acid | 7172 (852) | 7386 (847)
  Taurochenodeoxycholic acid | 1467 (204) | 1393 (195)
  Lithocholic acid | 74.02 (13.14) | 67.64 (14.64)
  Glycolithocholic acid | 165.3 (32.3) | 192.1 (57.8)
  Taurolithocholic acid | 21.66 (3.04) | 21.02 (4.55)
  Ursodeoxycholic acid | 116.5 (24.3) | 243.7 (159.7)
  Glycoursodeoxycholic acid | 415.5 (57.4) | 542.1 (181.9)
  Tauroursodeoxycholic acid | 19.79 (3.81) | 17.07 (3.33)
Statistical Analysis 1: Comparison: Polysorbate 80 vs Placebo; Test type: Equivalence — For each of 15 endogenous bile acid, simple one-way t-test to assess if endogenous bile acid AUC value is larger after polysorbate 80 than after placebo; p < 0.05, t-test, 1 sided

12. Secondary Outcome: Peak Plasma Concentration (Cmax) of Endogenous Bile Acids After Metformin
Description: For each of 15 endogenous bile acid, endogenous bile acid Cmax after metformin, compared to endogenous bile acid Cmax after placebo. Cmax units are concentration (i.e. ng/ml).
Time Frame: 0-10 hours
Measure: Mean (Standard Error); unit: ng/ml
Arm/Group | Metformin | Placebo
Number analyzed (Participants) | 12 | 12
ng/ml
  Cholic acid | 109.6 (40.5) | 123.8 (51.0)
  Glycocholic acid | 149.8 (37.5) | 263.9 (44.8)
  Taurocholic acid | 28.58 (6.20) | 67.64 (12.96)
  Deoxycholic acid | 234.0 (44.9) | 199.7 (28.6)
  Glycodeoxycholic acid | 338.1 (61.1) | 375.7 (50.9)
  Taurodeoxycholic acid | 49.66 (8.07) | 86.14 (16.50)
  Chenodeoxycholic acid | 2782 (451) | 2982 (359)
  Glycochenodeoxycholic acid | 1338 (267) | 1667 (234)
  Taurochenodeoxycholic acid | 192.9 (32.9) | 349.8 (69.7)
  Lithocholic acid | 10.88 (1.62) | 9.400 (2.040)
  Glycolithocholic acid | 36.20 (6.84) | 43.31 (12.76)
  Taurolithocholic acid | 4.020 (0.610) | 6.150 (1.800)
  Ursodeoxycholic acid | 65.54 (39.40) | 41.60 (24.98)
  Glycoursodeoxycholic acid | 121.5 (42.6) | 118.0 (38.3)
  Tauroursodeoxycholic acid | 3.350 (0.420) | 5.010 (0.930)
Statistical Analysis 1: Comparison: Metformin vs Placebo; Test type: Equivalence — For each of 15 endogenous bile acid, simple one-way t-test to assess if endogenous bile acid Cmax value is reduced after metformin than after placebo; p < 0.05, t-test, 1 sided

13. Secondary Outcome: Area-Under-the-Curve (AUC) of Endogenous Bile Acids After Metformin
Description: For each of 15 endogenous bile acid, endogenous bile acid AUC after metformin, compared to endogenous bile acid AUC after placebo. AUC units are concentration x time (i.e. ng/ml x h).
Time Frame: 0-10 hours
Measure: Mean (Standard Error); unit: ng/ml x h
Arm/Group | Metformin | Placebo
Number analyzed (Participants) | 12 | 12
ng/ml x h
  Cholic acid | 212.0 (46.3) | 259.7 (64.6)
  Glycocholic acid | 678.5 (131.4) | 1053 (187)
  Taurocholic acid | 126.5 (30.2) | 248.1 (39.5)
  Deoxycholic acid | 1366 (314) | 1222 (158)
  Glycodeoxycholic acid | 1618 (269) | 1507 (200)
  Taurodeoxycholic acid | 233.3 (36.9) | 329.3 (53.1)
  Chenodeoxycholic acid | 5290 (353) | 5552 (471)
  Glycochenodeoxycholic acid | 6499 (1122) | 7386 (847)
  Taurochenodeoxycholic acid | 879.8 (132.5) | 1393 (195)
  Lithocholic acid | 70.10 (10.74) | 67.64 (14.64)
  Glycolithocholic acid | 164.3 (30.3) | 192.1 (57.8)
  Taurolithocholic acid | 17.39 (3.00) | 21.02 (4.55)
  Ursodeoxycholic acid | 283.5 (168.9) | 243.7 (159.7)
  Glycoursodeoxycholic acid | 625.9 (220.8) | 542.1 (181.9)
  Tauroursodeoxycholic acid | 15.03 (3.17) | 17.07 (3.33)
Statistical Analysis 1: Comparison: Metformin vs Placebo; Test type: Equivalence — For each of 15 endogenous bile acid, simple one-way t-test to assess if endogenous bile acid AUC value is reduced after metformin than after placebo; p < 0.05, t-test, 1 sided

14. Secondary Outcome: Peak Plasma Concentration (Cmax) of Endogenous Bile Acids After Polysorbate 80
Description: For each of 15 endogenous bile acid, endogenous bile acid Cmax after polysorbate 80, compared to endogenous bile acid Cmax after placebo. Cmax units are concentration (i.e. ng/ml).
Time Frame: 0-10 hours
Measure: Mean (Standard Error); unit: ng/ml
Arm/Group | Polysorbate 80 | Placebo
Number analyzed (Participants) | 12 | 12
ng/ml
  Cholic acid | 91.16 (21.41) | 123.8 (51.0)
  Glycocholic acid | 291.3 (35.5) | 263.9 (44.8)
  Taurocholic acid | 77.80 (10.81) | 67.64 (12.96)
  Deoxycholic acid | 270.9 (49.4) | 199.7 (28.6)
  Glycodeoxycholic acid | 385.7 (43.5) | 375.7 (50.9)
  Taurodeoxycholic acid | 92.58 (13.42) | 86.14 (16.50)
  Chenodeoxycholic acid | 3049 (280) | 2982 (359)
  Glycochenodeoxycholic acid | 1396 (175) | 1667 (234)
  Taurochenodeoxycholic acid | 332.6 (47.4) | 349.8 (69.7)
  Lithocholic acid | 12.35 (2.59) | 9.400 (2.040)
  Glycolithocholic acid | 36.68 (7.81) | 43.31 (12.76)
  Taurolithocholic acid | 5.510 (0.760) | 6.150 (1.800)
  Ursodeoxycholic acid | 27.89 (5.30) | 41.60 (24.98)
  Glycoursodeoxycholic acid | 86.27 (12.40) | 118.0 (38.3)
  Tauroursodeoxycholic acid | 5.360 (0.770) | 5.010 (0.930)
Statistical Analysis 1: Comparison: Polysorbate 80 vs Placebo; Test type: Equivalence — For each of 15 endogenous bile acid, simple one-way t-test to assess if endogenous bile acid Cmax value is larger after polysorbate 80 than after placebo; p < 0.05, t-test, 1 sided

ADVERSE EVENTS:
Time Frame: Approximately 6 weeks, which is the duration of participant participation in the study.
Groups:
- Metformin: Participants took 500 mg metformin for 6 days. On day 7, participants were administered the cocktail, which included 80 mg pravastatin and 250 mg CDCA.
- Polysorbate 80: Participants took 400 mg polysorbate 80 b.i.d. for 6 days. On day 7, participants were administered the cocktail, which included 500 mg valacyclovir, 250 mg CDCA, 20 mg enalaprilat, and 400 mg polysorbate 80.
- Placebo: Participants took one placebo b.i.d. for 6 days. On day 7, participants were administered the cocktail, which included 500 mg valacyclovir, 250 mg CDCA, 20 mg enalaprilat, and 80 mg pravastatin.
Arm/Group | Metformin | Polysorbate 80 | Placebo
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/12 | 0/13
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/12 | 0/13
Other Adverse Events (participants affected / at risk) | 8/13 | 2/12 | 4/13
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Metformin (N=13) | Polysorbate 80 (N=12) | Placebo (N=13)
Diarrhea (Gastrointestinal disorders) | 3 | 0 | 1
Lightheaded and vision tunneling (Nervous system disorders) | 0 | 0 | 1
Elevated liver function tests (Hepatobiliary disorders) | 1 | 0 | 1
Vasovasgal syncope (Nervous system disorders) | 0 | 0 | 1
Easy bowel movement (Gastrointestinal disorders) | 2 | 1 | 0
Stomach discomfort and uneasiness (Gastrointestinal disorders) | 1 | 0 | 0
Stomach ache/pain (Gastrointestinal disorders) | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 3 | 0 | 0
Headache (Nervous system disorders) | 2 | 0 | 0
Stomach cramping (Gastrointestinal disorders) | 1 | 0 | 0
Mildly elevated alanine aminotransferase (Hepatobiliary disorders) | 1 | 0 | 0
GI issues (tightness and not feeling regular) (Gastrointestinal disorders) | 1 | 0 | 0
Fatigue (General disorders) | 1 | 0 | 0
Abdominal tightness (Gastrointestinal disorders) | 1 | 0 | 0
Wet/runny stool (Gastrointestinal disorders) | 1 | 0 | 0
Itchy rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-01-23): https://cdn.clinicaltrials.gov/large-docs/71/NCT04640571/Prot_SAP_000.pdf